CLINICAL TRIAL: NCT04505345
Title: Virtual Reality Cognitive Training in Individuals With Alcohol Use Disorder Undergoing Residential Treatment: A Randomized Controlled Trial
Brief Title: Virtual Reality Cognitive Training in Alcohol Use Disorder
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Universidade Lusófona de Humanidades e Tecnologias (Other)
Collaborators: Casa de Saúde do Telhal - Instituto São João de Deus, Portugal. (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SLB_AUD02
Record Dates: First submitted 2020-08-03; First posted 2020-08-10 (Actual); Last update posted 2023-05-11 (Actual); Status verified 2023-05

CONDITIONS: Cognitive Function; Feasibility

STUDY DESIGN:
Intervention Model Description: The individuals will be distributed by two groups: experimental and control. The experimental group consists of treatment with virtual reality cognitive training and the control group of treatment-as-usual.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Virtual reality cognitive training (Experimental): Virtual reality cognitive training consists of a behavioral intervention of 10 sessions of training using virtual reality exercises depicting daily life activities from the Systemic Lisbon Battery aiming cognitive impairments.
  Interventions: Behavioral: Cognitive training using the Systemic Lisbon Battery
- Treatment-as-usual (Other): Treatment-as-usual for alcohol use disorder (AUD) in our partner institution, a therapeutic community for rehabilitation of AUD, is conducted according to the Minnesota Model requiring alcohol abstinence.
  Interventions: Behavioral: Treatment-as-usual

INTERVENTIONS:
Behavioral: Cognitive training using the Systemic Lisbon Battery — The Systemic Lisbon Battery comprises exercises for cognitive rehabilitation developed to describe diverse activities of daily living.
  Arms: Virtual reality cognitive training
Behavioral: Treatment-as-usual — Treatment as usual for alcohol use disorder from Casa de Saúde do Telhal is delivered according to the Minnesota Model.
  Arms: Treatment-as-usual

SUMMARY:
This study aims to test the feasibility of using exercises in virtual reality for cognitive training of patients with alcohol use disorder undergoing residential treatment.

DETAILED DESCRIPTION:
Alcohol use disorder has been associated with diverse physical and mental morbidities. Among the main consequences of chronic and excessive alcohol use are cognitive and executive deficits. Some of these deficits may be reversed, with improvements in specific cognitive and executive domains, with behavioral approaches consisting in cognitive training. The advent of computer-based interventions may leverage these improvements, but RCTs on the use of digital interactive-based intervention are still scarce.

The aim consists in exploring whether a cognitive training approach using virtual reality exercises based on activities of daily living is feasible for improving cognitive function in patients with alcohol use disorder undergoing residential treatment.

The method consists in a two-arm randomized controlled trial with individuals recovering from alcohol use disorder in a therapeutic community that will be assigned to an experimental and a control group. The experimental group consists of virtual reality-based cognitive training whereas the control group of treatment-as-usual. A comprehensive neuropsychological battery of tests will be used consisting in tests for global cognition, executive functions, and specific tests form memory, attention and cognitive flexibility. The AB design will involve a baseline assessment before intervention and post-intervention assessment.

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years old
* Without history of psychiatric or neurological disorders
* Attending the inpatient program for rehabilitation of alcohol use disorder

Exclusion Criteria:

* Psychosis episode during the intervention
* Withdrawal from the inpatient program for rehabilitation of alcohol use disorder

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2017-09-30 (Actual); Primary Completion 2018-09-30 (Actual); Study Completion 2024-07-30 (Estimated)

PRIMARY OUTCOMES:
Executive functions | 5 weeks
  Executive functions are a set of higher order cognitive functions that control goal directed behavior. Executive functions in this study are assessed using the Frontal Assessment Battery that evaluates six constructs: conceptualization, mental flexibility, programming, sensitivity to interference, inhibitory control, and environmental autonomy. This study focuses on the total score that is calculated from sum of scores to each of the six dimensions of the test, in which higher scores describe better test performance.
Cognitive flexibility | 5 weeks
  Cognitive flexibility describes the ability to switch between different tasks. Cognitive flexibility in this study is assessed using the Wisconsin Card Sorting Test that evaluates strategic planning, abstract thinking, and capacity for perseveration and the ability to use environmental feedback. This test in this study is scored on six performance parameters: Number of trials administered; number of total errors; number of perseverative errors; number of trials to complete first category; failure to maintain set; and number of conceptual level responses. Higher scores in these dimensions reflect poorer test performance, except for the number of conceptual level responses.
Global cognition | 5 weeks
  Global cognition is assessed using the Montreal Cognitive Assessment that is a cognitive screening test that consists of 11 items assessing cognitive domains such as visuospatial orientation, naming, memory, attention, language, abstraction, evocation and orientation. This study focuses on the total score that is calculated from the sum of scores to each dimension of the test, in which higher scores reflect better test performance.

CONTACTS AND LOCATIONS:
Overall Officials: Pedro Gamito, PhD, Principal Investigator — University Lusófona
Locations (1):
- Casa de Saúde do Telhal, Sintra, Portugal

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Gamito P, Oliveira J, Matias M, Cunha E, Brito R, Lopes PF, Deus A. Virtual Reality Cognitive Training Among Individuals With Alcohol Use Disorder Undergoing Residential Treatment: Pilot Randomized Controlled Trial. J Med Internet Res. 2021 Jan 29;23(1):e18482. doi: 10.2196/18482. PMID 33512329